CLINICAL TRIAL: NCT07080346
Title: Upadacitinib for Refractory Behcet's Syndrome: a Prospective Pilot Open-label Study
Brief Title: Upadacitinib for Refractory Behcet's Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Liu Tian (Other)
Responsible Party: Sponsor-Investigator, Liu Tian, associate professor, Peking University People's Hospital
Organization: Peking University People's Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PKU People's Hospital UPA
Record Dates: First submitted 2025-07-15; First posted 2025-07-23 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-07

CONDITIONS: Behcet Syndrome
Keywords: Behcet syndrome; Upadacitinib
MeSH Terms: conditions — Behcet Syndrome | interventions — upadacitinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treated with upadacitinib (Experimental): Refractory BS patients were treated with upadacitinib.
  Interventions: Drug: Upadacitinib 15 MG

INTERVENTIONS:
Drug: Upadacitinib 15 MG — All the BS patients discontinued other biologic agents and received oral upadacitinib treatment at a dose of 15mg per day with background glucocorticoids and immunosuppressants for 48 weeks. All the patients will be followed up prospectively for 48 weeks.

SUMMARY:
Behçet's syndrome (BS) is a systemic autoimmune vasculitis that can affect multiple organs, including the skin, eyes, and vascular system. Refractory BS poses significant treatment challenges, necessitating novel therapeutic approaches. Upadacitinib, a selective JAK1 inhibitor within the JAK-STAT pathway, has shown promise in modulating immune responses. This study aims to evaluate the efficacy and safety of upadacitinib in patients with refractory BS.

DETAILED DESCRIPTION:
This multicenter, single-arm study investigates the efficacy and safety of upadacitinib (15 mg once daily) in refractory Behçet's syndrome (BS) patients. Adult patients had active BS with inadequate response to glucocorticoids and at least two conventional immunosuppressants or biologics over six months. Prior biologics were discontinued, and upadacitinib was added to ongoing glucocorticoids and immunosuppressants for 48 weeks. Clinical symptoms (oral/genital ulcers, skin lesions, uveitis), inflammatory markers (CRP, ESR), and medication usage were monitored. Adverse events were recorded to assess safety.

ELIGIBILITY:
Inclusion Criteria:

* • Male or female aged 18-70 years at time of screening.

  * Diagnosis of Behcet's syndrome (according to the International Criteria for Behçet's Disease) for ≥3 months before screening.
  * Active Behcet's syndrome at time of screening (BDCAF≥2).
  * Resistant to glucocorticoids, at least two traditional immunosuppressants (one of which must have been cyclophosphamide or mycophenolate mofetil) or biological agents (one of which must have been a TNF-α inhibitor or a JAK inhibitor) for at least 6 months.
  * Given their written informed consent to participate in the trial and expected to be able to adhere to the study visit schedule and other protocol requirements.

Exclusion Criteria:

* High-dose glucocorticoid (>1mg/kg/d) usage within 1 month.
* Severe comorbidities: including heart failure (≥ grade III NYHA), renal insufficiency (creatinine clearance ≤30 ml/min), hepatic insufficiency (serum ALT or AST >3 times the ULN, or total bilirubin >ULN for the central laboratory conducting the test). Other severe, progressive or uncontrolled hematologic, gastrointestinal, endocrine, pulmonary, cardiac, neurologic, or cerebral disease (including demyelinating diseases such as multiple sclerosis).
* Known allergies, hypersensitivity, or intolerance to Baricitinib or its excipients.
* Had a severe infection (including, but not limited to hepatitis, pneumonia, sepsis, or pyelonephritis); had been hospitalized for an infection; or had been treated with IV antibiotics for an infection, within 2 months prior to the first administration of study agent.
* Chest radiograph within 3 months prior to the first administration of study agent that showed an abnormality suggestive of a malignancy or current active infection, including tuberculosis.
* Infected with HIV (positive serology for HIV antibody) or hepatitis C (positive serology for Hep C antibody). If seropositive, consultation with a physician with expertise in the treatment of HIV or hepatitis C virus infection was recommended.
* Infected with hepatitis B virus. For patients who were not eligible for this study due to hepatitis B virus test results, consultation with a physician with expertise in the treatment of hepatitis B virus infection was recommended.
* Had any known malignancy or has a history of malignancy within the previous 5 years (with the exception of a nonmelanoma skin cancer that had been treated with no evidence of recurrence for ≥3 months before the first study agent administration or cervical neoplasia with surgical cure).
* Had uncontrolled psychiatric or emotional disorder, including a history of drug and alcohol abuse within the past 3 years that might prevent the successful completion of the study.
* Received, or was expected to receive, any live virus or bacterial vaccination within 3 months before the first administration of study agent, during the study, or within 4 months after the last administration of study agent. Had a BCG vaccination within 12 months of screening.
* Pregnancy, lactation or women of child-bearing potential (WCBP) unwilling to use medically approved contraception whilst receiving treatment and for 12 months after treatment has finished.
* Men whose partners are of child-bearing potential but who are unwilling to use appropriate medically approved contraception whilst receiving treatment and for 12 months after treatment has finished.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2024-01-25 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2025-07-08 (Actual)

PRIMARY OUTCOMES:
Patients getting improved condition | Week 24
  The primary endpoint was defined as the proportion(percent) of patients in the whole cohort getting improved condition by week 24. Improved condition was defined as BS-related manifestations resolved and no newly onset imaging/endoscopic findings observed.

SECONDARY OUTCOMES:
Changes of Behcet's Disease Current Activity Form (BDCAF) score of patients | Week 24 and week 48
  The clinical manifestation of patients were recorded during the follow-up. The disease activity of patients was accessed by Behcet's Disease Current Activity Form (BDCAF) score and the BDCAF scores (Range: 0~12, higher scores mean higher disease activity) at week 24, week 48 and the baseline scores were compared.
Changes of C-reactive protein | Week 24 and week 48
  Blood samples were collected from all patients and the concentration of C-reactive protein (mg/L) were recorded. C-reactive protein at 24 weeks, 48 weeks and the baseline were compared.
Changes of erythrocyte sedimentation rate | Week 24 and week 48
  Blood samples were collected from all patients and the erythrocyte sedimentation rates (mm/h) were recorded. Erythrocyte sedimentation rates at 24 weeks, 48 weeks and the baseline were compared.
Changes of dosage of glucocorticoids from baseline | Week 24 and week 48
  The dosage of glucocorticoids (mg/day) of all patients were recorded during the follow-up. The dosage of glucocorticoids at 24 weeks, 48 weeks and the baseline were compared.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Rheumatology and Immunology, Peking University People's Hospital, Beijing, Beijing Municipality, China